CLINICAL TRIAL: NCT01736189
Title: Assessment of Clinical Effectiveness and Safety of Adalimumab and High Dose Methotrexate in Routine Clinical Practice (Combo Study; Adalimumab With High Dose MTX)
Brief Title: Assessment of Clinical Effectiveness and Safety of Adalimumab and High Dose Methotrexate in Routine Clinical Practice
Status: Completed | Type: Observational
Sponsor: AbbVie (prior sponsor, Abbott) (Industry)
Responsible Party: Sponsor
Organization: AbbVie (Industry)
Other Study IDs: P13-684
Record Dates: First submitted 2012-11-27; First posted 2012-11-29 (Estimated); Results first posted 2019-07-02 (Actual); Last update posted 2019-07-02 (Actual); Status verified 2019-06

CONDITIONS: Rheumatoid Arthritis
Keywords: Rheumatoid arthritis; Methotrexate
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — Adalimumab

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Participants treated with adalimumab: 40 mg adalimumab via subcutaneous (SC) injection every other week (eow) for 104 weeks
  Interventions: Drug: Adalimumab

INTERVENTIONS:
Drug: Adalimumab — Pre-filled syringe, administered by subcutaneous injection
  Other Names: Humira; ABT-D2E7

SUMMARY:
This was a single-arm, multicenter, open label, prospective cohort study (post-marketing observational study) to determine the effectiveness and safety of adalimumab in combination with high-dose methotrexate (≥12 mg/week) in participants with rheumatoid arthritis in a routine clinical setting in Japan.

DETAILED DESCRIPTION:
Study assessments occurred at baseline, Week 12, Week 24, Week 52, Week 76, and Week 104. Most participants received 40 mg of adalimumab every other week during the study. Two participants started at 40 mg of adalimumab every other week, and increased to 80 mg every other week. A few participants had a different dose regimen: 40 mg every three weeks for 3 participants; 40 mg every four weeks for 1 participant; and 40 mg every other week with a switch to 50 mg every three weeks for 4 subjects.

ELIGIBILITY:
Inclusion Criteria:

The participants of this study were rheumatoid arthritis (RA) patients for whom adalimumab was prescribed. They must have met the following conditions:

* Disease duration of RA ≤2 years
* Methotrexate (MTX) administration ≥3 months prior to starting adalimumab
* Dose of MTX ≥12mg/week
* Disease Activity Score 28 (DAS28)-C-reactive protein (CRP) score >3.2

Exclusion Criteria:

* Participants who had been previously treated with biologics (including tumor necrosis factor [TNF] inhibitors and others)

Ages: 16 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Participants with rheumatoid arthritis treated in a daily clinical setting, who received adalimumab (and high dose methotrexate [≥12 mg/week]), were observed prospectively.
Sampling Method: Non-Probability Sample
Enrollment: 346 (Actual)
Dates: Start 2012-10-11 (Actual); Primary Completion 2018-04-16 (Actual); Study Completion 2018-04-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: AbbVie Inc., Study Director — AbbVie

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Tanaka Y, Mimori T, Yamanaka H, Sunaga N, Morita K, Kimura J, Takeuchi T. Effectiveness, safety, and methotrexate dose-tapering pattern over two years of treatment with adalimumab and >/=12 mg/week methotrexate for early rheumatoid arthritis: Results of the HAWK postmarketing surveillance study in Japan. Mod Rheumatol. 2020 May;30(3):424-433. doi: 10.1080/14397595.2019.1639931. Epub 2019 Jul 22. PMID 31267801
- See also: Related Info — http://rxabbvie.com

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: All registered participants
Period: Overall Study
Arm/Group | Participants Treated With Adalimumab
Started | 346
Completed | 300
Not Completed | 46
Not completed — Violation of registration criteria | 41
Not completed — Protocol Violation | 4
Not completed — Criteria and protocol violations | 1

BASELINE CHARACTERISTICS:
Population: Safety analysis set
Arm/Group | Participants Treated With Adalimumab
Number analyzed (Participants) | 300
Age, Continuous [Mean (Standard Deviation); unit: years] | 54.1 (13.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 221
  Male | 79
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With a Disease Activity Score 28 (DAS28) Score of <2.6 at Week 52
Description: The Disease Activity Score 28 (DAS28) is a validated index of rheumatoid arthritis disease activity. Twenty-eight tender joint counts, 28 swollen joint counts, the erythrocyte sedimentation rate (ESR; mm/hr) or C-reactive protein (CRP; mg/dL) level, and the participant's assessment of global disease activity (on a visual analog scale [VAS] from 0 to 10 cm) are included in the DAS28 score. Scores on the DAS28 range from 0 to 10; higher scores indicate more disease activity. A DAS28 score >5.1 indicates high disease activity, a DAS28 score <3.2 indicates low disease activity, and a DAS28 score <2.6 indicates clinical remission.
Time Frame: At Week 52
Population: Efficacy analysis set: participants with evaluable DAS-28 data
Measure: Number; unit: percentage of participants
Arm/Group | Participants Treated With Adalimumab
Number analyzed (Participants) | 292
percentage of participants
  DAS28-4CRP | 77.1
  DAS28-4ESR | 61.1

2. Secondary Outcome: Percentage of Participants With a Clinical Disease Activity Index (CDAI) Score ≤ 2.8 at Week 104
Description: The Clinical Disease Activity Index (CDAI) is a composite index for assessing rheumatoid arthritis disease activity. Twenty-eight tender joint counts, 28 swollen joint counts, the participant's global assessment of disease activity (on a visual analog scale [VAS] from 0 to 10 cm), and a physician's global assessment of disease activity (measured on a VAS from 0 to 10 cm) are summed to yield the total score. The total CDAI score ranges from 0 to 78 with higher scores indicating higher disease activity. Remission is defined as a CDAI score ≤ 2.8.
Time Frame: At Week 104
Population: Efficacy analysis set: participants with evaluable data
Measure: Number; unit: percentage of participants
Arm/Group | Participants Treated With Adalimumab
Number analyzed (Participants) | 131
percentage of participants | 69.5

3. Secondary Outcome: Percentage of Participants With a Simplified Disease Activity Index (SDAI) Score ≤ 3.3 at Week 104
Description: The SDAI is a validated measure of rheumatoid arthritis disease activity. Twenty-eight tender joint counts, 28 swollen joint counts, global disease activity assessed by the participant on a visual analogue scale from 0 to 10 (cm), global disease activity assessed by an investigator on a visual analogue scale from 0 to 10 (cm), and serum levels of C-reactive protein (CRP; mg/dL) were included in the SDAI score. Scores on the SDAI range from 0 to 86. An SDAI score ≥26.1 indicates high disease activity, an SDAI score between 11.1 and 26.0 indicates moderate disease activity, an SDAI score between 3.4 and 11.0 indicates low disease activity, and an SDAI score ≤3.3 indicates clinical remission.
Time Frame: At Week 104
Population: Efficacy analysis set: participants with evaluable data
Measure: Number; unit: percentage of participants
Arm/Group | Participants Treated With Adalimumab
Number analyzed (Participants) | 128
percentage of participants | 73.4

4. Secondary Outcome: Percentage of Participants With a Health Assessment Questionnaire Disability Index (HAQ-DI) Score < 0.5 at Week 104
Description: The Health Assessment Questionnaire - Disability Index (HAQ-DI) is a self-reported assessment specific for rheumatoid arthritis. It consists of 20 questions referring to eight domains: dressing/grooming, arising, eating, walking, hygiene, reach, grip, and daily activities. Participants assessed their ability to do each task over the past week using the following response categories: without any difficulty (0); with some difficulty (1); with much difficulty (2); and unable to do (3). Scores on each task were summed and averaged to provide an overall score ranging from 0 to 3, where zero represents no disability and three very severe, high-dependency disability. HAQ remission indicating normal physical function is defined as HAQ-DI < 0.5.
Time Frame: At Week 104
Population: Efficacy analysis set: participants with evaluable data
Measure: Number; unit: percentage of participants
Arm/Group | Participants Treated With Adalimumab
Number analyzed (Participants) | 105
percentage of participants | 90.5

5. Secondary Outcome: Mean Change From Baseline in European Quality of Life-5 Dimensions Health Questionnaire (EQ-5D) Index Score at Week 104
Description: The European Quality of Life-5 Dimensions Health Questionnaire (EQ-5D) is a participant-answered questionnaire scoring 5 dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. For each dimension the participant is asked for a three-level assessment of their health on the current day: "no problems" (1), "some problems" (2), "extreme problems" (3). EQ-5D health states, defined by the EQ-5D descriptive system, are converted into a single summary index by applying a formula that essentially attaches values (also called QOL weights or QOL utilities) to each of the levels in each dimension. EQ-5D Summary Index values range from -0.11 (worst health state) to 1.00 (perfect health state). Positive numbers indicate improvement from baseline.
Time Frame: Baseline and Week 104
Population: Efficacy analysis set: participants with evaluable data
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Participants Treated With Adalimumab
Number analyzed (Participants) | 95
units on a scale | 0.2543 (0.1950)

6. Secondary Outcome: Percentage of Participants With a Change From Baseline of ≤ 1.0 in Van Der Heijde Modified Total Sharp Score (mTSS) at Week 104
Description: The van der Heijde modified Total Sharp Score (mTSS) is a measure of the level of joint damage. X-rays of hands and feet were taken at the visit. Joints were scored for erosions on a scale of 0 (no damage) to 5 (complete collapse) and joint space narrowing on a scale of 0 (no damage) to 4 (ankylosis or complete dislocation). Erosion scores and narrowing scores were added to obtain the mTSS (range = 0 [normal] to 398 [maximal disease]). An increase in mTSS from Baseline represents disease progression and/or joint worsening, no change represents halting of disease progression, and a decrease represents improvement.
Time Frame: Baseline and Week 104
Population: Efficacy analysis set: participants with evaluable data
Measure: Number; unit: percentage of participants
Arm/Group | Participants Treated With Adalimumab
Number analyzed (Participants) | 70
percentage of participants | 84.3

ADVERSE EVENTS:
Time Frame: Treatment-emergent adverse events (TEAEs) and serious adverse events (TESAEs) were collected from the time of study drug administration until the end of the study (up to 104 weeks).
Description: TEAEs and TESAEs are defined as any adverse event (AE) with an onset date that is after the first dose of study drug and were collected whether elicited or spontaneously reported by the participant.
Arm/Group | Participants Treated With Adalimumab
All-Cause Mortality (participants affected / at risk) | 0/300
Serious Adverse Events (participants affected / at risk) | 29/300
Other Adverse Events (participants affected / at risk) | 0/300
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Participants Treated With Adalimumab (N=300)
BRONCHOPULMONARY ASPERGILLOSIS (Infections and infestations) | 1 (1)
CELLULITIS (Infections and infestations) | 1 (1)
PNEUMONIA (Infections and infestations) | 1 (1)
PNEUMONIA CYTOMEGALOVIRAL (Infections and infestations) | 1 (1)
PNEUMONIA LEGIONELLA (Infections and infestations) | 1 (1)
PNEUMONIA PNEUMOCOCCAL (Infections and infestations) | 2 (2)
PNEUMONIA STREPTOCOCCAL (Infections and infestations) | 1 (1)
PNEUMOCYSTIS JIROVECII PNEUMONIA (Infections and infestations) | 4 (4)
BASAL CELL CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
COLON CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
DIFFUSE LARGE B-CELL LYMPHOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
OVARIAN CANCER METASTATIC (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
LUNG NEOPLASM MALIGNANT (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
PANCYTOPENIA (Blood and lymphatic system disorders) | 2 (2)
THROMBOCYTOPENIA (Blood and lymphatic system disorders) | 1 (1)
CEREBRAL HAEMORRHAGE (Nervous system disorders) | 1 (1)
MENINGITIS NONINFECTIVE (Nervous system disorders) | 1 (1)
VITREOUS HAEMORRHAGE (Eye disorders) | 1 (1)
INTERSTITIAL LUNG DISEASE (Respiratory, thoracic and mediastinal disorders) | 1 (1)
COLITIS (Gastrointestinal disorders) | 1 (1)
INGUINAL HERNIA (Gastrointestinal disorders) | 1 (1)
LIVER DISORDER (Hepatobiliary disorders) | 1 (1)
RASH (Skin and subcutaneous tissue disorders) | 1 (1)
URTICARIA (Skin and subcutaneous tissue disorders) | 1 (1)
SPONDYLOLISTHESIS (Musculoskeletal and connective tissue disorders) | 1 (1)
RENAL DISORDER (Renal and urinary disorders) | 1 (1)
RENAL IMPAIRMENT (Renal and urinary disorders) | 1 (1)
TUBULOINTERSTITIAL NEPHRITIS AND UVEITIS SYNDROME (Renal and urinary disorders) | 1 (1)
UTERINE HAEMORRHAGE (Reproductive system and breast disorders) | 1 (1)
BLOOD PRESSURE DECREASED (Investigations) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
AbbVie requests that any investigator or institution that plans on presenting/publishing results disclosure, provide written notification of their request 60 days prior to their presentation/publication. AbbVie requests that no presentation/publication will be instituted until 12 months after a study is completed, or after the first presentation/publication whichever occurs first. A delay may be proposed of a presentation/publication if AbbVie needs to secure patent or proprietary protection.

DOCUMENTS (2):
  • Study Protocol (2017-12-11): https://cdn.clinicaltrials.gov/large-docs/89/NCT01736189/Prot_000.pdf
  • Statistical Analysis Plan (2018-04-09): https://cdn.clinicaltrials.gov/large-docs/89/NCT01736189/SAP_001.pdf